CLINICAL TRIAL: NCT01747135
Title: Hydroxypropyl Beta Cyclodextrin for Niemann-Pick Type C1 Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vtesse, LLC, a Mallinckrodt Pharmaceuticals Company (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130001
Record Dates: First submitted 2012-12-08; First posted 2012-12-11 (Estimated); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Niemann-Pick Disease, Type C1
Keywords: 2-Hydroxypropyl-B-Cyclodextrin; Niemann-Pick Disease, Type C1; Neurodegeneration
MeSH Terms: conditions — Niemann-Pick Disease, Type C; Nerve Degeneration | interventions — 2-Hydroxypropyl-beta-cyclodextrin

ARMS (1):
- Open label (Experimental)
  Interventions: Drug: VTS-270

INTERVENTIONS:
Drug: VTS-270
  Other Names: 2-hydroxypropyl-beta-cyclodextrin

SUMMARY:
Background:

- Hydroxypropyl beta cyclodextrin (HPBCD) is being tested for a disease called Niemann-Pick disease type C1 (NPC1). NPC1 is a genetic disorder that results in gradual loss of nervous system function. Cholesterol and other fats have trouble moving out of the brain cells, which makes the cells work poorly and leads to symptoms. There is no treatment currently approved in the US for NPC1. Researchers want to test if it is safe to use HPBCD for NPC1. They want to see if it can help brain cells process cholesterol better.

Objectives:

- To test the safety and effectiveness of HPBCD for NPC1.

Eligibility:

- Individuals between 2 and 25 years of age who have been diagnosed with NPC1 and who have not already received HPBCD in an attempt to treat NPC1.

Design:

* Participants will be screened with a physical exam and medical history. They will provide blood and urine samples for screening. They will also have neurological tests, including tests of hearing, speech and movement.
* Participants will have a lumbar puncture (also called a spinal tap) every month to deliver the drug to the spinal fluid that surrounds the brain. The length of the trial will be determined by the safety and efficacy information that is obtained.
* Treatment will be monitored with frequent blood and urine tests, cerebral spinal fluid tests, hearing and neurological exams.

DETAILED DESCRIPTION:
Niemann-Pick disease type C (NPC) is a lethal, autosomal recessive, lysosomal storage disorder characterized by neurodegeneration in early childhood and death in adolescence. The causative genes NPC1 (about 95% of cases) and NPC2 (about 5% of cases) are involved in the intracellular trafficking of lipids and cholesterol. Mutations on either of these genes lead to progressive accumulation of unesterified cholesterol and other lipids in the central nervous system (CNS). The National Institutes of Health (NIH) Therapeutics for Rare and Neglected Diseases (TRND) program is developing 2-hydroxypropyl-Beta-cyclodextrin (HP-Beta-CD) for the treatment of patients with Niemann-Pick disease type C1 (NPC1) to slow progression of symptoms of the disease. In this Phase 1, non-randomized, open-label, single-center, study, we propose to administer HP-Beta-CD intrathecally via lumbar injection to drug naive cohorts of 3 patients at doses of 200 mg escalated to 300, 400 mg and 900 mg. Subsequent dose escalations may occur in increments of up to 300 mg. The objectives of this study are to assess the safety, tolerability, feasibility, and pharmacokinetics (PK) of intrathecally (IT) administered HP-Beta-CD to NPC1 patients, to determine an active dose of HP-Beta-CD as measured by changes in plasma 24-(S) hydroxycholesterol (24(S)-HC) concentration, and to evaluate the use of biomarkers and potential clinical outcomes of NPC1. All patients in the cohort will receive HP-Beta-CD (n = 3) once monthly for at least two doses, and the decision to dose-escalate will be based on safety and on biochemical data. Safety will be assessed by adverse events (AEs), audiologic evaluation, clinical laboratory tests, vital signs, physical examinations, chest X-rays and electrocardiograms (ECGs). Biochemical efficacy will be measured by change from baseline in plasma 24(S)-HC. PK will be assessed for plasma HP-Beta-CD.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Aged greater than or equal to 2 and less than or equal to 25 years old at time of enrollment, either gender and any ethnicity.
  2. Diagnosis of NPC1 based upon one of the following:

     1. Two NPC1 mutations;
     2. Positive filipin staining and at least one NPC1 mutation;
     3. Vertical supranuclear gaze palsy (VSNGP) in combination with either:

     i. One NPC1 mutation, or

     ii. Positive filipin staining and no Niemann-Pick Type 2 (NPC2) mutations.
  3. Patients with at least one neurological manifestation of NPC1. For example, but not limited to, hearing loss, vertical supranuclear gaze palsy, ataxia, dementia, dystonia, seizures, dysarthria, or dysphagia.
  4. Ability to travel to the National Institutes of Health Clinical Center (NIH CC) repeatedly for evaluation and follow-up.
  5. If taking miglustat, the patient must have been taking a constant dose of the medication for no less than 3 months prior to baseline evaluation and must be willing to maintain that dose level for the duration of the trial.
  6. Willing to discontinue all non-prescription supplements, with the exception of an age-appropriate multivitamin.
  7. Women of reproductive age must be willing to use an effective method of contraception for the duration of the trial.
  8. Willing to participate in all aspects of trial design including serial blood and cerebrospinal fluid (CSF) collections.

     EXCLUSION CRITERIA:

  <!-- -->

  1. Aged below 2 or above 25 years of age at enrollment in the trial.
  2. Subjects will be excluded if their weight would result in an endotoxin level that would exceed 0.2 EU/kg for either the saline or drug dosing.
  3. Severe manifestations of NPC1 that would interfere with the patient's ability to comply with the requirements of this protocol.
  4. Neurologically asymptomatic patients.
  5. Patients who have received any form of cyclodextrin in an attempt to treat NPC1. Treatment with another drug preparation for another medical indication that contains cyclodextrin as an excipient, will not exclude a patient.
  6. History of hypersensitivity reactions to cyclodextrin or components of the formulation.
  7. Pregnancy or breastfeeding at any time during the study.
  8. Patients with suspected infection of the CNS or any systemic infection.
  9. Spinal deformity that would impact the ability to perform a lumbar puncture
  10. Skin infection in the lumbar region
  11. Neutropenia, defined as an absolute neutrophil count (ANC) of less than 1,500.
  12. Thrombocytopenia (a platelet count of less than 75,000 per cubic millimeter).
  13. Evidence of disturbed circulation of CSF.
  14. Contraindication for anesthesia.
  15. Prior use of anticoagulants or history/presence of a bleeding disorder with increased risk of clinical bleeding or an international normalized ratio (INR) greater than 2.
  16. Patients with clinical evidence of acute liver disease having symptoms of jaundice or right upper quadrant pain.
  17. Presence of anemia defined as two standard deviations below normal for age and gender.
  18. For subjects 18 years of age and older, the epidermal growth factor receptor (eGFR) is automatically calculated and reported by the NIH CC laboratory utilizing the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) Creatinine 2009 equation. We will exclude subjects greater than or equal to 18 years of age if eGFR is less than or equal to 60 mL/min/1.73 m2. For subjects < 18

  12 years of age, we will utilize the national kidney disease education program (NKDEP) calculator (http://www.nkdep.nih.gov/lab-evaluation/gfr-calculators/children-conventional-unit.shtml). Results are reported as > 75 mL/min/1.73 m2 or lower. We will exclude subjects < 18 years of age if eGFR is less than or equal to 75 15 mL/min/1.73 m2

  19. Hematuria on a single urinalysis, as defined by the American Urological Association (AUA) as five or more red blood cells per high-power field (or > 25/micro L) on microscopic evaluation of urinary sediment from a properly collected urinalysis specimen. The patient will not be excluded if 2 subsequent urine specimens are negative for hematuria as defined by the AUA.

  20. Proteinuria (1+ protein on urinalysis) unless evaluated and classified as benign by patient s primary medical provider or by NIH nephrology consult or in the context of normal urine protein creatinine ratio and in the absence of clinical symptoms (edema, hypertension).

  21. Active pulmonary disease, oxygen requirement or clinically significant history of decreased blood oxygen saturation, pulmonary therapy, or requiring active suction.

  22. Patients unable to complete a behavioral audiologic evaluation including pure-tone threshold assessment (500 Hz to 8000 Hz) to monitor for ototoxicity and for whom otoacoustic emissions (OAEs) cannot be reliably obtained at baseline.

  23. Patients with ongoing seizures, that are not stable in frequency, type or duration over a 2 month period prior to enrollment, requiring change in dose of antiepileptic medication (other than adjustment for weight) over a 2 month period prior to enrollment, or requiring 3 or more antiepileptic medications to control seizures.

  24. Patients, who in the opinion of the investigators are unable to comply with the protocol or have specific health concerns that would potentially increase the risk of participation.

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2013-01; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
24-hydroxycholesterol Area under the curve | Days

SECONDARY OUTCOMES:
Hearing loss. | Year

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Mallinckrodt
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Publish in peer reviewed journal

REFERENCES:
- [Background] Aqul A, Liu B, Ramirez CM, Pieper AA, Estill SJ, Burns DK, Liu B, Repa JJ, Turley SD, Dietschy JM. Unesterified cholesterol accumulation in late endosomes/lysosomes causes neurodegeneration and is prevented by driving cholesterol export from this compartment. J Neurosci. 2011 Jun 22;31(25):9404-13. doi: 10.1523/JNEUROSCI.1317-11.2011. PMID 21697390
- [Background] Brewster ME, Loftsson T. Cyclodextrins as pharmaceutical solubilizers. Adv Drug Deliv Rev. 2007 Jul 30;59(7):645-66. doi: 10.1016/j.addr.2007.05.012. Epub 2007 May 29. PMID 17601630
- [Background] Chen FW, Li C, Ioannou YA. Cyclodextrin induces calcium-dependent lysosomal exocytosis. PLoS One. 2010 Nov 29;5(11):e15054. doi: 10.1371/journal.pone.0015054. PMID 21124786
- [Derived] Farmer C, Lewis M, Farhat N, Robbins KP, Joseph L, Albert OK, Bianconi S, Hoffmann A, Giserman-Kiss I, Alexander DM, Thurm A, Porter FD, Kravis EB. Convergent Validity of the Fine Motor, Speech, and Cognitive Domains of the 5-Domain Niemann-Pick Disease Type C Clinical Severity Scale. J Child Neurol. 2026 Jan;41(1):43-53. doi: 10.1177/08830738251346348. Epub 2025 Jun 17. PMID 40525490
- [Derived] Boenzi S, Catesini G, Sacchetti E, Tagliaferri F, Dionisi-Vici C, Deodato F. Comprehensive-targeted lipidomic analysis in Niemann-Pick C disease. Mol Genet Metab. 2021 Dec;134(4):337-343. doi: 10.1016/j.ymgme.2021.11.005. Epub 2021 Nov 16. PMID 34810067
- [Derived] Farmer CA, Thurm A, Farhat N, Bianconi S, Keener LA, Porter FD. Long-Term Neuropsychological Outcomes from an Open-Label Phase I/IIa Trial of 2-Hydroxypropyl-beta-Cyclodextrins (VTS-270) in Niemann-Pick Disease, Type C1. CNS Drugs. 2019 Jul;33(7):677-683. doi: 10.1007/s40263-019-00642-2. PMID 31187454
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2013-CH-0001.html